CLINICAL TRIAL: NCT00705991
Title: Validation of Thrombelastometry (ROTEM®)
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: StV 27-2007
Record Dates: First submitted 2008-01-17; First posted 2008-06-27 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2012-11

CONDITIONS: Coagulation
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: ROTEM

SUMMARY:
Das Hauptziele der Studie ist das ROTEM® zu validieren durch die Untersuchung von:

i) Reproduzierbarkeit von ROTEM® ii) Präzision der ROTEM®-Tests, sowie iii) der Zeitspanne, während derer die Ergebnisse in Zitrat-Blut reproduzierbar sind

Die durchzuführenden Tests sind FIBTEM, EXTEM, INTEM in ROTEM® um die Funktion der Thrombozyten während der Lagerungszeit zu untersuchen.

Nur Zitrat-Blut wird den Patienten abgenommen, die Reklazifikation findet kurz vor der Durchführen der Tests stattfinden, um so nahe wie möglich an der klinischen Praxis zu sein.

ELIGIBILITY:
Inclusion criteria: 1. Vorgesehen für einen elektiven Eingriff 2. Unterschriebene Einverständniserklärung

Exclusion criteria: 1. bekannte Tumorerkrankung oder Immunosupression, 2. bekannte Gerinnungsstörung 3. Antikoagulation 4. Behandlung mit Heparin über 3000 UI im Sinne der Thrombose-Prophylaxe hinaus 5. Gebrauch von Acetylsalicylsäure innerhalb der letzten 5 Tage 6. Gebrauch von NSRA innerhalb der letzten 24 Stunden 7. bekannte Niereninsuffizienz oder eine Plasmakonzentration von Kreatinin grösser 120 Mm, oder Lebererkrankungen oder einer Plasmakonzentration von ASAT (> 50 U/l) oder ALAT (> 50 U/l).

8. Patienten / Patientinnen und Probanden / Probandinnen die der Deutschen Sprache nicht mächtig sind.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy Patients
Sampling Method: Non-Probability Sample
Dates: Start 2008-01; Study Completion 2008-10

CONTACTS AND LOCATIONS:
Overall Officials: Donat R Spahn, Prof MD, Principal Investigator — University Hospital Zurich, Division of Anaesthesiology
Locations (1):
- Zurich, Switzerland